CLINICAL TRIAL: NCT06931236
Title: Clinical Efficacy and Mechanism of Repetitive Transcranial Magnetic Stimulation Based on dlPFC in the Intervention of Generalized Anxiety Disorder With Insomnia: An Open-label Study
Brief Title: Clinical Efficacy and Mechanism of rTMS Based on dlPFC in the Intervention of Generalized Anxiety Disorder With Insomnia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yanghua Tian (Other)
Responsible Party: Sponsor-Investigator, Yanghua Tian, Vice President of Anhui Medical University, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-TMS-GADIS
Record Dates: First submitted 2025-03-30; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Generalized Anxiety Disorder (GAD); Insomnia; Repetitive Transcranial Magnetic Stimulation (rTMS)
Keywords: generalized anxiety disorder; insomnia; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Generalized Anxiety Disorder; Sleep Initiation and Maintenance Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- real stimulation (Active Comparator): Stimulation was performed using a figure 8-shaped focal coil attached to a MagPro 100 magnetic stimulator (MagVenture, Copenhagen, Denmark). All patients received 1 Hz (10 s trains, 1 s inter-train interval, 1,360 pulses per session) rTMS treatment once daily on weekdays for 2 consecutive weeks. rTMS was delivered over the right DLPFC (F4 electrode site according to the International 10-20 EEG system) at 100% of the resting motor threshold (RMT).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- sham stimulation (Sham Comparator): sham rTMS is carried out as the coil is turned away from the skull at 90°.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive transcranial magnetic stimulation (rTMS) can noninvasively modulate cortical activity by delivering a sequence of magnetic pulses.
  Arms: real stimulation
Device: Sham Repetitive Transcranial Magnetic Stimulation — Sham tDCS was delivered using the same protocol and current intensity, but it is carried out as the coil is turned away from the skull at 90°.
  Arms: sham stimulation

SUMMARY:
To investigate the intervention effect of Repetitive Transcranial Magnetic Stimulation (rTMS) on insomnia symptoms of generalized anxiety disorder patients.

DETAILED DESCRIPTION:
Stimulation was performed using a figure 8-shaped focal coil attached to a MagPro 100 magnetic stimulator (MagVenture, Copenhagen, Denmark). All patients received 1 Hz (10 s trains, 1 s inter-train interval, 1,360 pulses per session) rTMS treatment once daily on weekdays for 2 consecutive weeks. rTMS was delivered over the right DLPFC (F4 electrode site according to the International 10-20 EEG system) at 100% of the resting motor threshold (RMT) . To determine the RMT, stimulus intensity was gradually increased until 5 out of 10 trials elicited motor evoked potentials with peak-to-peak amplitudes over 50 μV in the contralateral abductor pollicis brevis muscle. Adverse events attributed to rTMS were documented and reported. All participants received a pre-treatment assessment with the PSQI, HAMA, and HAMD. We used the PSQI to measure sleep quality, as well as HAMA and HAMD to assess participant's anxious and depressive states. Likewise, the PSQI was measured post-treatment (upon completion of the final treatment session) and at 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. age between 15 and 65 years;
2. clinically diagnosed with anxiety according to the Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V);
3. no previous application of any insomnia pharmacological therapy for at least one week before baseline visit.

Exclusion Criteria:

1. current or history of serious brain and body diseases;
2. current or history of schizophrenia, behavioral problems, post-traumatic stress disorder, mania, obsessive-compulsive disorder, and social phobia;
3. substance abuse or other comorbid psychological diseases.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
subjective sleep quality assessed by the PSQI | before and after 10-day intervention and at 1-month follow-up
  The Pittsburgh Sleep Quality Index (PSQI) consist of 18 items divided into 7 dimensions, such as sleep duration, sleep efficiency, sleep disorders and daytime dysfunction. The PSQI total score ranges from 0 to 21, the higher the score indicates the more worse sleep quality.
subjective sleep quality assessed by the ISI | before and after 10-day intervention and at 1-month follow-up
  The Insomnia Severity Index (ISI) is a 7-item scale to measure insomnia symptoms, where each item is rated on a scale from 0 to 4. The ISI total score ranges from 0 to 28, The higher the score indicates the more worse sleep quality.
emotional symptoms assessed by the HAMA | before and after 10-day intervention and at 1-month follow-up
  The HAMA is a 14-item scale to measure the severity of anxiety symptoms, where each item is rated on a scale from 0 to 4. The HAMA total score ranges from 0 to 56, with lower scores indicating less anxiety symptoms.

SECONDARY OUTCOMES:
emotional symptoms assessed by the HAMD | before and after 10-day intervention and at 1-month follow-up
  The HAMD is a clinic ian-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China